CLINICAL TRIAL: NCT00001028
Title: A Randomized, Comparative, Prospective Study of Monthly Aerosolized Pentamidine and Thrice Weekly Dapsone for Prophylaxis Against PCP in HIV-Infected Patients Who Are Intolerant to Trimethoprim and/or Sulfonamides
Brief Title: A Study of Pentamidine Plus Dapsone in the Prevention of Pneumocystis Carinii Pneumonia (PCP) in HIV-Infected Patients Who Cannot Take Trimethoprim or Sulfonamides
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Jacobus Pharmaceutical (Industry); Fujisawa Pharmaceutical Co (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CPCRA 013; 11565 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Pentamidine; Dapsone; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Pentamidine; Dapsone

INTERVENTIONS:
Drug: Pentamidine isethionate
Drug: Dapsone

SUMMARY:
To compare the safety and efficacy of aerosolized pentamidine and dapsone in the prevention of Pneumocystis carinii pneumonia (PCP) in high-risk HIV-infected patients who are intolerant to trimethoprim and/or sulfonamides.

Both aerosolized pentamidine and dapsone have been shown to prevent PCP, but both drugs cause side effects. This study attempts to determine which drug is more efficacious as prophylaxis against PCP in patients who cannot tolerate trimethoprim/sulfamethoxazole.

DETAILED DESCRIPTION:
Both aerosolized pentamidine and dapsone have been shown to prevent PCP, but both drugs cause side effects. This study attempts to determine which drug is more efficacious as prophylaxis against PCP in patients who cannot tolerate trimethoprim/sulfamethoxazole.

Patients are evenly divided between two treatment arms to receive either aerosolized pentamidine every 4 weeks or dapsone orally three times weekly. Follow-up data is collected every 3 months, and patients are clinically evaluated every 6 months. Patients who develop PCP or a severe or persistent study drug toxicity may be switched to the alternative study drug at the clinician's discretion. Average duration of follow-up is 2 years.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 count <= 200 cells/mm3 or <= 15 percent of total lymphocytes OR a history of prior PCP.
* History of intolerance to trimethoprim and/or sulfonamides.
* No active pneumocystosis. Patient or guardian must sign informed consent. Pregnant patients are eligible at the clinician's discretion. Patients who do not meet required laboratory values may be eligible at the discretion of the clinician.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Any medication with potential anti-PCP activity.

Patients with the following prior conditions are excluded:

* Treatment-limiting reaction to pentamidine or dapsone.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Study Completion 1994-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: El-Sadr W, Study Chair; Luskin-Hawk R, Study Chair
Locations (14):
- United States (14):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Wishard Hosp / Indiana Univ Hosp, Indianapolis, Indiana
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] el-Sadr W, Wentworth D, Dehlinger M, Larntz K. Design and implementation of a community-based trial for prophylaxis for P. carinii pneumonia (PCP). Int Conf AIDS. 1993 Jun 6-11;9(1):79 (abstract no WS-B36-2)